CLINICAL TRIAL: NCT02517736
Title: Study Multicentre Evaluating the Effectiveness and Toxicity Sorafenib (Nexavar®) in Adult Patients With Uveal Melanoma and Metastatic Dissemination
Acronym: O-Mel-Sora
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-067
Record Dates: First submitted 2015-08-05; First posted 2015-08-07 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sorafenib at a dose of 800 mg / day (Experimental)
  Interventions: Drug: Sorafenib at a dose of 800 mg / day

INTERVENTIONS:
Drug: Sorafenib at a dose of 800 mg / day

SUMMARY:
The objective of the study is to determine the efficacy and toxicity of sorafenib in metastatic uveal melanoma.

The main objective is to determine the non-tumor progression rate 24 weeks after initiation of treatment with sorafenib at a dose of 800 mg / day

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years old suffering from uveal melanoma with metastasis
* At least one measurable metastases by more than 10 mm acoording to Response Evaluation Criteria in Solid Tumors (RECIST)
* At least 28 days from the previous treatment (systemic or major surgery)
* Performance Index (WHO ≤ 2 or ≥ 70% Karnofsky)
* Weight loss compared to pre morbid weight <20% in the last 12 months
* White blood cells at least 3000 / mm 3, polynuclear neutrophils less than 1500 / mm3, platelets at least 100,000 / mm3, hemoglobin at least 9.0 g / dl
* Total Bilirubin ≤1.5 x upper limit of normal (ULN) (or less than or equal to 2.5 in liver metastasis), ASAT and ALAT ≤ 2.5 x ULN (or ≤ 5 in liver metastasis) Serum Creatinine (calculated using the cockcroft-Gault method) ≤ 1.5 x ULN, Amylase and lipase <1.5 x ULN
* prothrombin rate and international normalized ratio (INR) or activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN. Possibility of using low molecular weight heparin in place of anti vitamin K treatment
* higher life expectancy than or equal to 3 months
* Negative pregnancy test for women of childbearing age and using a method of contraception during treatment
* No one benefiting from a Social Security scheme
* Informed consent and signed by the patient or his legal representative

Exclusion Criteria:

* • Patient who received more than 2 lines of treatment (chemotherapy or immunotherapy), whatever the indication

  * Major surgery (excluding the possible diagnostic biopsy) or radiation therapy in the 4 weeks preceding the inclusion
  * single liver metastasis treatable by surgery
  * active peptic ulcer, uncontrolled
  * Other progressive malignancy or during treatment (except basal cell carcinoma)
  * Cardiac arrhythmias requiring anti-arrhythmic (excluding beta-blockers or digoxin for chronic atrial fibrillation), active or ischemic coronary disease (myocardial infarction within the last 6 months), or heart failure> New York Heart Association (NYHA) class II
  * Bacterial or fungal infection active (grade> 2 Common Toxicity Criteria for Adverse Effects (CTCAE) v4.03)
  * known HIV infection or chronic hepatitis B or C
  * cerebral or meningeal tumor metastasis (symptomatic or asymptomatic)
  * epileptic disease requiring anti-epileptic taken
  * Previous history of organ transplantation or peripheral stem cells
  * Patient kidney dialysis
  * Concomitant treatment with cytochrome P450 3A4 (CYP3A4) inducers such as rifampin, St. John's wort, phenytoin, carbamazepine, phenobarbital and dexamethasone
  * Prior therapy with bevacizumab or other targeted therapy
  * Known or suspected allergy to sorafenib
  * Any unstable chronic illness can jeopardize patient safety or its compliance
  * Women pregnant or lactating
  * coagulopathy
  * Uncontrolled hypertension
  * Inability to swallow
  * Failure to submit to medical monitoring of the trial due to geographical, social or psychic
  * Persons deprived of liberty or under supervision
  * Patient refusing ambulatory care
  * Patient simultaneously participating in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2012-02 (Actual); Primary Completion 2015-01-13 (Actual); Study Completion 2015-01-13 (Actual)

PRIMARY OUTCOMES:
non-tumor progression rate | 24 weeks after initiation of treatment
  with sorafenib at a dose of 800 mg / day

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'ophtalmologie, CHU de Caen, Caen, France